CLINICAL TRIAL: NCT03917745
Title: E-health Intervention in Women With Pregnancy Distress: a Randomized Controlled Trial
Brief Title: E-health Intervention in Women With Pregnancy Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Responsible Party: Principal Investigator, prof.dr. Victor J Pop, Principal Investigator, Tilburg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50-54300-98-244
Record Dates: First submitted 2019-04-03; First posted 2019-04-17 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy Distress
Keywords: anxiety; depression; eHealth; mindfulness; pregnancy distress
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The study is part of a large longitudinal cohort study among pregnant women. The study targets a specific subgroup of pregnant women with symptoms of psychological distress (depression and anxiety). Women who score above cut off on the Edinburgh Depression Scale (EDS) and Tilburg Pregnancy Distress Scale (TPDS) at 12 weeks of gestation, will be randomly allocated to the intervention or control group. Women in the intervention group will be contacted and invited to participate in the mindfulness-based intervention, which consists of 8 weeks of internet mindfulness training. The control group will receive care as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHealth mindfulness intervention group (Experimental): 8 weeks of internet mindfulness training
  Interventions: Behavioral: eHealth mindfulness intervention
- Control group (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: eHealth mindfulness intervention — The web-based intervention consists of eight sessions including psycho-education about the mechanisms of stress, coping and relaxation, especially related to pregnancy, practicing mindfulness skills (i.e. mindful breathing, mindful moving, observing and letting-go of thoughts and emotions with a non-judgmental attitude), sharing experiences, and doing home assignments. The sessions have been developed specifically for pregnant women and acknowledge pregnancy-related distress. An online coach will review questions and home assignments of the participants. Women will start the training at 16 weeks gestation.
  Other Names: Ontspannen zwanger
  Arms: eHealth mindfulness intervention group

SUMMARY:
The study aims to reduce the levels of distress (depression and anxiety) during pregnancy. The study investigates the effectiveness of an eHealth pregnancy distress-reducing mindfulness training in women with pregnancy distress.

DETAILED DESCRIPTION:
During pregnancy, women are at risk for mental health problems: up to 20% present with distress symptoms (depression and/or anxiety). Apart from the adverse effects on the woman herself, pregnancy distress negatively affects pregnancy outcome, infant health, postpartum mother-child interaction and child development.

Mindfulness-based interventions are a type of intervention that is increasingly being used to treat symptoms of stress, anxiety and depression. They are cheap and accessible to the whole population.

Current study aims to examine the effectiveness of a mindfulness training to reduce distress during pregnancy. Women who score above cut off on the Edinburgh Depression Scale (EDS) and Tilburg Pregnancy Distress Scale (TPDS) at 12 weeks of gestation, will be randomly allocated to the intervention or control group. Women in the intervention group will be contacted and invited to participate in the mindfulness-based intervention, which consists of 8 weeks of internet mindfulness training. The control group will receive care as usual.

The primary outcome of the study is: Does the mindfulness internet training "Ontspannen zwanger", offered during pregnancy, reduce pregnancy distress, compared to care as usual? The secondary outcome is: Does the mindfulness internet training result in better mindfulness skills?

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (18+y) who have their first antenatal visit < 12 weeks;
* Score above cut off on the Edinburgh Depression Scale (EDS) and Tilburg Pregnancy Distress Scale (TPDS) at 12 weeks of gestation;
* Dutch-speaking or understanding Dutch.

Exclusion Criteria:

* Gemelli pregnancy (or higher order pregnancy);
* Known endocrine disorder before pregnancy (diabetes-I, Rheumatoid arthritis);
* Severe psychiatric disease (schizophrenia, borderline or bipolar disorder);
* HIV;
* Drug or alcohol addiction problems;
* Any other disease resulting in treatment with drugs that are potentially adverse for the fetus and need careful follow-up during pregnancy;
* No access to the internet.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Difference between the intervention group en the control group, measured at 28 weeks (after the intervention).
  Measured by the 10-item Edinburgh Depression Scale (EDS). The EDS is the most widely used self-rating scale to assess depressive symptoms in the perinatal period. It consists of ten items and three sub-scales: anhedonia, anxiety and depression. The questionnaire has been validated in Dutch pregnant women. The EDS total score ranges from 0 to 30, with higher scores indicating more depressive symptoms.

SECONDARY OUTCOMES:
Negative Affect | Difference between the intervention group en the control group, measured at 28 weeks (after the intervention).
  Measured by a subscale of the Tilburg Pregnancy Distress Scale (TPDS): Negative Affect, which consists of 10 items. The TPDS has been validated among Dutch pregnant women and it is a reliable measure to assess pregnancy-related emotional distress. The total score ranges from 0 to 30, with higher scores indicating more emotional distress symptoms.

OTHER OUTCOMES:
Mindfulness skills | Measured in the intervention group, the difference between 16 weeks (before the intervention) and 28 weeks (after the intervention).
  Measured by three facets of the Five Facet Mindfulness Questionnaire Short Form (FFMQ-3-SF): acting with awareness, non-judging and non-reacting, which consists of 15 items. The validity of the measure is established and indices of internal reliability were found to be adequate. The total score ranges from 0 to 60, with higher scores indicating better mindfulness skills.
Rumination | Measured in the intervention group, the difference between 16 weeks (before the intervention) and 28 weeks (after the intervention).
  Measured by the Rumination-Reflection Questionnaire (RRQ), which consists of 12 items and is a validated and reliable instrument. The score ranges from 0 to 48, with higher scores indicating more rumination.
Self compassion | Measured in the intervention group, the difference between 16 weeks (before the intervention) and 28 weeks (after the intervention).
  Measured by the Self Compassion Scale Short Form (SCS-SF), which consists of 12 items, and is a validated and reliable measure. The total score ranges from 0 to 72, with higher scores indicating higher self compassion.

CONTACTS AND LOCATIONS:
Locations (1):
- Tilburg University, Tilburg, Netherlands

REFERENCES:
- [Derived] Hulsbosch LP, Potharst ES, Schwabe I, Boekhorst MGBM, Pop VJM, Nyklicek I. Online mindfulness-based intervention for women with pregnancy distress: A randomized controlled trial. J Affect Disord. 2023 Jul 1;332:262-272. doi: 10.1016/j.jad.2023.04.009. Epub 2023 Apr 12. PMID 37054897
- [Derived] Hulsbosch LP, Nyklicek I, Potharst ES, Meems M, Boekhorst MGBM, Pop VJM. Online mindfulness-based intervention for women with pregnancy distress: design of a randomized controlled trial. BMC Pregnancy Childbirth. 2020 Mar 13;20(1):159. doi: 10.1186/s12884-020-2843-0. PMID 32169030